CLINICAL TRIAL: NCT05624073
Title: Comparison of Blind Tracheal Intubation Through the Air-QTM Blocker and the LarySealTM Pro Laryngeal Mask Airways in Anesthetized Paralyzed Adult Patients Undergoing Elective Ophthalmic Operations
Brief Title: Blind Tracheal Intubation Through Supraglottic Airway Devices
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Ali Abdelhaleem Abdelrahman, Anesthesia lecturer M.D., Cairo University
Other Study IDs: EH-2022
Record Dates: First submitted 2022-11-13; First posted 2022-11-21 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Respiration and the Airways With Laryngeal Masks
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Air-QTM Blocker: GA (n=35): Air-Q Blocker TM will be used as a conduit for blind endotracheal intubation.
  Interventions: Device: LarySealTM Pro
- LarySealTM Pro Laryngeal Mask: GL (n=35): Laryseal TM Pro will be used as a conduit for blind endotracheal intubation.
  Interventions: Device: Air-QTM Blocker

INTERVENTIONS:
Device: Air-QTM Blocker — The Air-QTM Blocker (Cookgas LLC, Mercury Medical, Clearwater, FL, USA) is a SAD that is intended for use as a primary airway seal and an aid for tracheal intubation in situations of anticipated or unanticipated difficult airways. Its design includes a large airway tube inner diameter, a short airway tube length, and a tethered, removable standard 15mm circuit adapter. These features enable direct insertion of larger tracheal tubes up to 7.5 and 8.5mm inner diameters for Air-Q sizes 3.5 and 4.5 respectively (according to body weight; size 3.5: 50-70Kg, size 4.5:70-100Kg). In addition to the soft blocker channel (guide tube) that acts as a conduit for placing medical devices such as NG (Nasogastric) or Blocker tubes. NG tubes are used to decompress and suction the stomach. Standard NG tubes up to 18 Fr. are suitable for all Air-Q Blocker sizes
  Groups: LarySealTM Pro Laryngeal Mask
Device: LarySealTM Pro — The LarysealTM Pro is the new generation mask for safe and effective airway management, as it could reduce the risk of aspiration by the integrated suction catheter port to allow effective removal of fluids and gastric contents. So that, it could be a promising airway device as its symmetrical cuff and tube contoured to match the oropharyngeal anatomy for quick and easy first time insertion success. It could be applied in both routine and advanced airway management for patients with a higher risk of a difficult airway, unexpected intubation difficulties, beside to airway control during anesthesia. It was presented in the clinical market in: sizes 3, 4 and 5 (according to the body weight; size 3: 30-50Kg, size 4: 50-70 Kg, and size 5:70-100Kg) that can accept larger tracheal tube up to 7.5 and 8mm inner diameter respectively with maximum suction catheter size of 16 Fr. Both devices accommodated standard conventional endotracheal tubes for intubation.
  Groups: Air-QTM Blocker

SUMMARY:
Tracheal intubation is considered the gold standard for protecting the airway. As the supraglottic airway devices (SADs) could be inserted without laryngoscopy, so that SADs with different designs and safety issues could be used to manage difficult airways in anesthesia and emergency medicine with continuous patient oxygenation &ventilation, less hemodynamic stress response and less postoperative complications. These advantages encourage the use of a proper SAD as a conduit for endotracheal intubation in stressful conditions. This study will be carried out to compare the Air-QTM Blocker and LarysealTM Pro for blind tracheal intubation during elective ophthalmic surgeries under general anesthesia. Intubation through SAD can be performed using a fiber-optic bronchoscope or blindly. Blind intubation is meaning that the tube is inserted through SAD without direct visualization of the airway. Success rate of blind intubation ranges between 15% and 97%, mostly depending on the type of used SAD, patient characteristics and operator skills. The availability of blind intubation through SAD is important in cases of difficult intubation (either anticipated or unanticipated) especially if fiber-optic is not available, so that SAD will be convenient for untrained personnel.

DETAILED DESCRIPTION:
The laryseal pro could provide rapid and secure airway management and improve patient safety with gastric access reducing the risk of pulmonary aspiration, in addition to speeding up the ETT tube placement with a unique guide system, beside to integrated fenestrated flap that protects from blockage with minimal increase in flow resistance, and elevates the epiglottis for easy, trauma-free ETT tube or bronchoscope insertion. According to the manufacturer: all these features of laryseal pro allow quick easy first time insertion success. As, the laryseal pro is being of shorter breathing tube and smaller cuff in comparison to Air-Q Blocker, so the laryseal pro is expecting to be more amazing than the Air-Q Blocker especially for the new trainers regarding the total insertion time of the endotracheal tube and success rate. Jatin et al. 2021reported that Air-Q Intubating Laryngeal Airway resulted in significantly more success rate and ease of intubation as compared to Ambu Aura Gain. Andrzej et al. 2018 stated that success rate of blind intubation through Air-Q was 75% when compared to 80% in I-gel group. In contrary, there are limited studies available in literature on blind tracheal intubation through the laryseal pro.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-55 years old.
2. ASA I&II.
3. Both sexes.
4. El-Ganzouri Airway Score < or =2

Exclusion Criteria:

1. History of upper respiratory tract infections.
2. History of obstructive sleep apnea (OSA) or STOP Bang-Score > 4.
3. Potentially full stomach (trauma, morbid obesity BMI> 35 Kg/m2, pregnancy, history of gastric regurgitation and heart burn).
4. Esophageal reflux (hiatus hernia).
5. Coagulation disorders.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Eligible subjects of both sexes will be consecutively enrolled and randomly allocated to LarysealTM Pro group or Air-QTM Blocker group through an online randomization program (http://www.randomizer.org) with an allocation ratio of 1:1.
  GL (n=35): Laryseal TM Pro will be used as a conduit for blind endotracheal intubation.
  GA (n=35): Air-Q Blocker TM will be used as a conduit for blind endotracheal intubation.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-12-17 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Total insertion time (seconds) | 200 seconds
  Total insertion time (seconds): insertion time (seconds) of the SAD is the time needed for correct SAD placement &started when SAD touched teeth to the first recorded rectangular capnogram curve with satisfactory bilateral chest expansion + insertion time of the endotracheal tube through the SAD (seconds) is the time in seconds from insertion of the endotracheal tube blindly until capnographic confirmation.

CONTACTS AND LOCATIONS:
Overall Officials: Reham Ali Abdelhaleem Abdelrahman, M.D., Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Department of Anesthesia, Surgical ICU, and Pain Management, Cairo
  - Reham Ali Abdelhaleem Abdelrahman, Cairo